CLINICAL TRIAL: NCT05117047
Title: Long-term Survival Analysis of Robotic, Laparoscopic and Open Liver Resection for Hepatocellular Carcinoma in BCLC Stage 0-A: A Prospective Cohort Study With Matched Comparison
Brief Title: A Long-term Survival Analysis of Different Surgical Method in Early Hepatocellular Carcinoma
Status: Completed | Type: Observational
Sponsor: Chen Xiaoping (Other)
Responsible Party: Sponsor-Investigator, Chen Xiaoping, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: C201501
Record Dates: First submitted 2021-11-03; First posted 2021-11-11 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Long-term Effects of Cancer Treatment
MeSH Terms: interventions — Hepatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- robot-assisted liver resection: In this study, the investigators included all HCC patients with BCLC stage 0-A (n=1669) who underwent hepatectomy over an 1 ½ year study period, and divided them into three study cohorts according to the operations they received. These were consecutive patients who met the inclusion criteria of the study. 71 HCC patients were included in robotic liver resection cohort.
  Interventions: Procedure: liver resection
- laparoscopic liver resection: In this study, the investigators included all HCC patients with BCLC stage 0-A (n=1669) who underwent hepatectomy over an 1 ½ year study period, and divided them into three study cohorts according to the operations they received. These were consecutive patients who met the inclusion criteria of the study. 141 HCC patients were included in laparoscopic liver resection cohort.
  Interventions: Procedure: liver resection
- open liver resection: In this study, the investigators included all HCC patients with BCLC stage 0-A (n=1669) who underwent hepatectomy over an 1 ½ year study period, and divided them into three study cohorts according to the operations they received. These were consecutive patients who met the inclusion criteria of the study. 157 HCC patients were included in open liver resection cohort.
  Interventions: Procedure: liver resection

INTERVENTIONS:
Procedure: liver resection — After adequate periods of follow-up, the long-term oncological outcomes of the three different surgical approaches were compared, providing a higher level of evidence using a non-randomized comparative study based on propensity score matching (PSM) analysis.

SUMMARY:
The investigators established three prospective cohorts of patients with BCLC stage 0-A HCC, based on different surgical approaches (open, laparoscopic and robotic). After 5 years of follow-up, the investigators used propensity score matching (PSM) to reduce selection bias and then compared the long-term oncological outcomes of the three different surgical approaches, which might provide high-level evidence in non-randomized observational studies.

DETAILED DESCRIPTION:
In this study, three prospective cohorts of patients with BCLC stage 0-A HCC, underwent complete liver resection using different surgical approaches (OLR, LLR, and RALR), were established. After adequate periods of follow-up, the long-term oncological outcomes of the three different surgical approaches were compared, providing a higher level of evidence using a non-randomized comparative study based on propensity score matching (PSM) analysis.

ELIGIBILITY:
Inclusion Criteria:

* All HCC patients in BCLC stage 0-A underwent liver resection in hepatic surgery center, Tongji hospital, Tongji Medical College, Huazhong University of Science and Technology. The inclusion criteria were as follows: 14- 75 years old

Exclusion Criteria:

* with any history of malignant tumors; with treatment of ablation, TACE or TKI history before liver resection.

Ages: 14 Years to 75 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 1669 cases underwent liver resection from July 1st 2015 to June 30th 2017 in Hepatic Surgery Center, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, including 186 RALR, 527 LLR, and 956 OLR. Among these patients, there were 102, 333, and 669 HCC patients, respectively. Ten patients were excluded due to missing data or follow-up. Finally, 369 HCC patients in the early stages were included in the analysis. After PSM, 168 patients were matched and there were 56 patients in each group
Sampling Method: Non-Probability Sample
Enrollment: 369 (Actual)
Dates: Start 2015-02-14 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 14/02/2015-30/06/2021
  The primary outcomes of this study included long-term oncological outcomes of OS
Disease free Survival | 14/02/2015-30/06/2021
  The primary outcomes of this study included long-term oncological outcomes of DFS

SECONDARY OUTCOMES:
postoperative complications | 14/02/2015-30/06/2021
  Postoperative morbidity and mortality were assessed according to the Clavien-Dindo classification
Textbook Outcome in liver surgery (TOLS) | 14/02/2015-30/06/2021
  Textbook Outcome in liver surgery (TOLS), was defined as the absence of intraoperative incidents of grade 2 or higher, postoperative bile leak grade B or C, severe postoperative complications, readmission within 30 days after discharge, in-hospital mortality, and the presence of R0 resection margin.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoping Chen, Dr, Study Chair — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China